CLINICAL TRIAL: NCT05660447
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled, Study on the Use of Rho-Kinase Inhibitor to Reduce Ore Prevent Proliferative Vitreoretinopathy (PVR) in Eyes With Rhegmatogenous Retinal Detachment (RRD) at High Risk of PVR
Brief Title: A Multi-Center Study on the Use of Rho-Kinase Inhibitor to Reduce or Prevent PVR in RRD Eyes at High Risk for PVR
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jason Hsu, MD, Co-Director, Retina Research; Associate Professor, Sidney Kimmel Medical College at Thomas Jefferson University, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB #2022-77
Record Dates: First submitted 2022-12-03; First posted 2022-12-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Rhegmatogenous Retinal Detachment; Proliferative Vitreoretinopathy
Keywords: retinal detachment; rhegmatogenous; proliferative vitreoretinopathy; rho kinase; netarsudil; rhopressa
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment; Hereditary Sensory and Autonomic Neuropathies | interventions — netarsudil; Ophthalmic Solutions; Glycerol; Hypromellose Derivatives; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Netarsudil 0.02% (Experimental): For the study arm: one drop of rho-kinase (ROCK) inhibitor in the vitrectomized eye, once daily in the evening starting on postoperative day 1 after RRD repair surgery, till post-operative day 56
  Interventions: Drug: Netarsudil 0.02% Ophthalmic Solution [RHOPRESSA]
- Artificial tears (Placebo Comparator): Patients enrolled in the control group will receive a placebo (one drop of artificial tears) once daily in the evening starting on postoperative day 1 after RRD repair surgery, till post-operative day 56
  Interventions: Drug: Glycerin 0.2%/Hypromellose 0.2%/Peg 1%/Soln,Oph,Ud

INTERVENTIONS:
Drug: Netarsudil 0.02% Ophthalmic Solution [RHOPRESSA] — One drop of rho-kinase (ROCK) inhibitor in the vitrectomized eye, once daily in the evening starting on postoperative day 1 after RRD repair surgery, till post-operative day 56
  Other Names: Rhopressa
  Arms: Netarsudil 0.02%
Drug: Glycerin 0.2%/Hypromellose 0.2%/Peg 1%/Soln,Oph,Ud — Patients enrolled in the control group will receive a placebo (one drop of artificial tears) once daily in the evening starting on postoperative day 1 after RRD repair surgery, till post-operative day 56
  Other Names: Geri-Care Artificial Tears
  Arms: Artificial tears

SUMMARY:
The purpose of this study is to determine if a drug called netarsudil is safe and able to prevent the development of scar tissue after retinal detachment repair. Patients eligible for this study are those diagnosed with a rhegmatogenous retinal detachment deemed at high risk for scar tissue formation (a process called 'proliferative vitreoretinopathy').

ELIGIBILITY:
Inclusion Criteria:

A patient must meet the following criteria to be eligible for inclusion in the study:

1. Diagnosed with primary RRD at high risk for PVR development. Specifically, the enrolled eye must include at least 1 but no more than 3 high risk features, which are designated as follows: multiple retinal breaks (3 or more); detachments involving two or more quadrants of the retina; duration of detachment > 3 weeks; vitreous hemorrhage; and choroidal detachment.
2. Consents to surgical repair with pars plana vitrectomy with or without scleral buckling
3. Willing and able to comply with clinic visits and study-related procedures
4. Able to provide a signed informed consent

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Age < 18 years
2. Presence of PVR grade B or worse (as defined by the revised Retina Society PVR classification system) at time of surgical repair
3. Primary RRD repair is primary laser demarcation, primary cryotherapy, pneumatic retinopexy, or scleral buckling procedure alone.
4. Primary use of silicone oil or retinectomy during surgical repair
5. Prior incisional ocular surgery other than cataract extraction
6. History of or concurrent ruptured globe, intraocular foreign body, diabetic retinopathy, retinal vein occlusion, exudative age-related macular degeneration, macular hole, epiretinal membrane, sickle cell disease, uveitis or intraocular infectious disease
7. Not willing or unable to comply with clinic visits and study-related procedures
8. Unable to provide a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Single surgery anatomic success (retinal re-attachment) rate | Six months
  Successful retinal re-attachment after the primary surgery without requiring additional surgical interventions.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed on ophthalmic examination at all time points. | Six months
  Adverse events of interest include endophthalmitis, intraocular inflammation, or retinal tear/detachment.
The number of participants with evidence of grade C proliferative vitreoretinopathy (PVR) on retinal examination. | Six months
  PVR Grade C is defined by preretinal or subretinal retinal membrane, including a retinal star fold
The number of participants with an epiretinal membrane as assessed on ocular examination or optical coherence tomography imaging | Six months
  Epiretinal membrane is defined as preretinal membrane overlying the macula.
Change from baseline in visual acuity (Snellen) wearing habitual correction. | Six months
  Visual acuity will be measured using a typical Snellen chart.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Wills Eye Physicians-Mid Atlantic Retina, Wills Eye Hospital
Locations (1):
- Wills Eye Physicians - Mid Atlantic Retina, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Townes-Anderson E, Wang J, Halasz E, Sugino I, Pitler A, Whitehead I, Zarbin M. Fasudil, a Clinically Used ROCK Inhibitor, Stabilizes Rod Photoreceptor Synapses after Retinal Detachment. Transl Vis Sci Technol. 2017 Jun 20;6(3):22. doi: 10.1167/tvst.6.3.22. eCollection 2017 Jun. PMID 28660097
- [Background] Halasz E, Townes-Anderson E, Zarbin MA. Improving outcomes in retinal detachment: the potential role of rho-kinase inhibitors. Curr Opin Ophthalmol. 2020 May;31(3):192-198. doi: 10.1097/ICU.0000000000000658. PMID 32235252